CLINICAL TRIAL: NCT04183868
Title: Comparative Effects of Empagliflozin Versus Glimepiride After 26-weeks of Treatment Add on Metformin on Myocardial Metabolic Rate of Glucose Estimated Through 18FDG-PET in Patients With Type 2 Diabetes
Brief Title: Effects of empagliFlozin on myocardIal metabOlic Rate of glucosE Estimated Through 18FDG PET (FIORE Study)
Acronym: FIORE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Catanzaro (Other)
Responsible Party: Principal Investigator, Elena Succurro, Associate Professor in Internal Medicine, University of Catanzaro
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2016.43
Record Dates: First submitted 2019-11-11; First posted 2019-12-03 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Type 2 Diabetes; Cardiovascular Risk Factor
Keywords: Empagliflozin; Type 2 diabetes; Myocardial glucose uptake; Cardiovascular risk
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin; glimepiride

STUDY DESIGN:
Intervention Model Description: 52-weeks, single-center, prospective, controlled, randomized, open-label, two parallel group and switch, active-comparator.
  13 subjects with T2DM, poorly controlled on metformin monotherapy, and without a history of ischemic heart disease, will be treated with empagliflozin for 26 weeks and will be compared with a group of 13 subjects with T2DM, poorly controlled on metformin monotherapy, and without a history of ischemic heart disease, treated with glimepiride (both in addition to metformin) for 26 weeks. At the end of 26 weeks of treatment, subjects belonging to the first group will be shifted to glimepiride therapy, while subjects belonging to the second group will be shifted to empagliflozin treatment for 26 weeks. All subjects, then, will control themselves.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

ARMS (2):
- Empagliflozin (Experimental): Eligible patients (meeting all inclusion criteria) will be randomized to receive empagliflozin in addition to existing metformin background therapy (daily dose of ≥1.500 mg, which has to remain unchanged throughout the study) for 26 weeks.
  At the end of 26 weeks of treatment, subjects belonging to empagliflozin arm will be shifted to glimepiride treatment.
  Interventions: Drug: Empagliflozin 10 MG
- Glimepiride (Active Comparator): Eligible patients will be randomized to receive glimepiride (starting dose: 2 mg daily) treatment arm, can undergo to up-titration of glimepiride to a maximum of 6 mg/day, if they experience fasting plasma glucose (FPG) levels > 112 mg/dl (6,2 mmol/l) at scheduled visit at 6th week or at any later scheduled visit.
  Whereas, glimepiride-treated patients experiencing recurrent hypoglycemic episodes should down-titrate glimepiride to a dose, considered as appropriate by Investigator.
  Hypoglycemic events are defined as symptoms suggestive of low blood glucose confirmed by self monitored blood glucose (SMBG) < 56 mg/dl (3,1 mmol/l).
  Severe hypoglycemia is defined as any hypoglycemic episode requiring the assistance of another party for recovery.
  At the end of 26 weeks of treatment, subjects belonging to glimepiride arm will be shifted to treatment with empagliflozin for 26 weeks.
  Interventions: Drug: Glimepiride 2 mg

INTERVENTIONS:
Drug: Empagliflozin 10 MG — 10 mg tablet daily
  Other Names: Jardiance
  Arms: Empagliflozin
Drug: Glimepiride 2 mg — starting dose: 2 mg tablet daily, 1 mg for lunch and 1 mg for dinner, can undergo to up-titration of glimepiride to a maximum of 6 mg daily
  Other Names: Solosa; Amaryl
  Arms: Glimepiride

SUMMARY:
Diabetes is an independent risk factor for ischemic heart disease (CAD) and heart failure, and cardiovascular diseases are the main cause of mortality and morbidity in patients with diabetes. Recent studies on cardiovascular outcomes have shown that type 2 sodium glucose co-transporter (SGLT-2i) inhibitors are not only effective in improving glycometabolic control, but are also able to reduce major CV events (MACE) and hospitalization for heart failure. However, it is still unclear whether the beneficial CV effects of treatment with SGLT2i are due to indirect mechanisms such as reduction in blood pressure, improvement of vascular stiffness, reduction in body weight and visceral adiposity, reduction in uricemia or whether they have effects direct on the heart. Recently, it was shown that in nondiabetic porcine model with heart failure, the treatment with empagliflozin was associated with a switch of myocardial fuel utilization from glucose uptake toward uptake of ketone bodies and free fatty acid, thereby improving myocardial energetics, enhancing LV systolic function, and ameliorating adverse LV remodeling.

It is not known whether empagliflozin treatment is able to modify the heart's energy metabolism even in humans.

In this study we hypothesize that empagliflozin may determine beneficial CV effects reducing myocardial metabolic rate of glucose assessed by hyperinsulinemic euglycemic clamp 18F-FDG PET scans in patients with type 2 diabetes.

This is a single-center, prospective, controlled, randomized, open-label, two parallel group and switch, active-comparator study that evaluates the comparative effects of 26 weeks of treatment with empagliflozin versus glimepiride add on metformin on myocardial metabolic rate of glucose estimated through 18F-FGD-PET scan in patients with type 2 diabetes without a history of coronary heart disease. At the end of 26 weeks of treatment, subjects belonging to the first group will be shifted to glimepiride therapy, while subjects belonging to the second group will be shifted to empagliflozin treatment for 26 weeks. All subjects, then, will control themselves.

DETAILED DESCRIPTION:
Diabetes mellitus type 2 (T2DM) is the most common metabolic disease and its prevalence is rapidly increasing. T2DM is a chronic disease that affects over 451 million people in the world and this number is expected to increase over the years and it is estimated that in 2045 there will be in the world over 693 million patients with T2DM. Diabetes is an independent risk factor for ischemic heart disease (CAD), stroke and peripheral artery disease and cardiovascular diseases are the main cause of mortality and morbidity in patients with diabetes. It is estimated that subjects with T2DM have a risk of cardiovascular events same as those of non-diabetic subjects with a previous cardiovascular event and several epidemiological studies have reported that the incidence of fatal and nonfatal coronary events in patients with T2DM is 1.5 to 3-4 times higher than non-diabetics of the same age.

Many studies showed that, in diabetic subjects, improved plasma glucose is associated with a reduction in microvascular complications. Instead, is not completely shown that a reduction of plasma glucose result in a reduction of cardiovascular events. In fact, although it was noted that, in subjects with T2DM, good control glyco-metabolic is associated with modest cardiovascular benefits in the long term, however, the intensive treatment hypoglycemic agent or the use of antidiabetic drugs is often associated with adverse events cardiovascular.

Recently, it was approved for the treatment of T2DM a new class of drugs, inhibitors of sodium glucose cotransporter type 2 (SGLT-2), that work by blocking the renal glucose reabsorption, causing glycosuria. SGLT-2 inhibitors have a good safety profile, are effective in reducing HbA1c regardless of the duration of diabetes and the degree of beta-cell dysfunction and insulin resistance and exhibit a low risk of hypoglycemia. In addition, the loss of glucose renal induced by SGLT2 inhibitors is associated with modest weight loss and reduction in blood pressure. Pre clinical studies showed that SGLT2 inhibitors, through a reduction in glucose toxicity, determine an improvement in insulin resistance liver and muscle and a restoration of first and second phase insulin secretion. The improvement of β-cell function and insulin sensitivity, assessed by indexes derived from OGTT, was obtained in subjects with T2DM, even after a single dose of empagliflozin, selective SGLT2 inhibitor. There are few data on the changes in insulin sensitivity, assessed by hyperinsulinemic euglycemic clamp, and insulin secretion, estimated by intravenous glucose test tolerance (IVGTT), induced by SGLT2 inhibitor. It was shown that, in subjects with T2DM at high cardiovascular risk, treatment with empagliflozin in addition to standard therapy was associated with a significant reduction of the composite cardiovascular endpoint, consisting of cardiovascular death, non-fatal myocardial infarction and non-fatal stroke, compared to placebo. In addition, treatment with empagliflozin in addition to standard therapy determined in a significant reduction in cardiovascular mortality, mortality from all causes and hospitalization for heart failure compared to placebo. It is not completely known the mechanism through which treatment with empagliflozin is associated to an improvement of cardiovascular outcomes. Growing evidences suggest that empagliflozin performs positive cardiovascular effects through a reduction in blood pressure, an improvement in arterial stiffness, a reduction in body weight and visceral adiposity. Recently, it was shown that in nondiabetic porcine model with heart failure, the treatment with empagliflozin was associated with a switch of myocardial fuel utilization from glucose uptake toward uptake of ketone bodies and free fatty acid, thereby improving myocardial energetics, enhancing LV systolic function, and ameliorating adverse LV remodeling.

Myocardial positron emission tomography (PET) with 18F-Fluorodeoxyglucose (18F-FDG), a widely used glucose analogue, in combination with the euglycemic-hyperinsulinemic clamp is considered the gold standard to measure myocardial metabolic rate of glucose under standardized experimental conditions. In this study we hypothesize that empagliflozin may determine beneficial cardiovascular effects reducing myocardial metabolic rate of glucose assessed by hyperinsulinemic euglycemic clamp 18F-FDG PET scans in patients with type 2 diabetes with no history of coronary heart disease, compared to treatment with glimepiride, both add on metformin.

Study design

13 subjects with T2DM, poorly controlled on metformin monotherapy, and without a history of ischemic heart disease, will be treated with empagliflozin for 26 weeks and will be compared with a group of 13 subjects with T2DM, poorly controlled on metformin monotherapy, and without a history of ischemic heart disease, treated with glimepiride (both in addition to metformin) for 26 weeks. At the end of 26 weeks of treatment, subjects belonging to the first group will be shifted to glimepiride therapy, while subjects belonging to the second group will be shifted to empagliflozin treatment for 26 weeks. All subjects, then, will control themselves.

Schematic overview of the study timeline

Visit 1 Screening (week -1): Clinical examination, vital signs (systolic and diastolic blood pressure and pulse), anthropometric measures, HbA1c, FPG, haematology and biochemistry, pro-BNP, high sensitivity C-reactive protein (hsCRP), troponin T, renal function, albumin/creatinine ratio (ACR), evaluation criteria for inclusion and exclusion, electrocardiogram (ECG), echocardiogram, Holter ECG.

Visit 2 Randomization (week 0 baseline): Hyperinsulinemic euglycemic clamp combined with 18F-FDG PET. Assignment two treatment arms randomly with ratio of 1: 1. Beginning of treatment with empagliflozin 10 mg/day in one arm and the other glimepiride.

Visit 3 (week 4): Clinical examination, security monitoring (systolic and diastolic blood pressure), hypoglycemia and adverse events evaluation

Visit 4 (week 8): Clinical examination, security monitoring (ECG (assessment of P Wave, QRS Complex, QT Interval), systolic and diastolic blood pressure), hypoglycemia and adverse events evaluation

Visit 5 (week 12): Clinical examination, security monitoring, hypoglycemia and adverse events evaluation

Visit 6 (week 26): Clinical examination, vital signs (systolic and diastolic blood pressure and pulse), anthropometric measures, haematology and biochemistry, pro-BNP, high sensitivity C-reactive protein (hsCRP), troponin T, renal function, ACR, ECG, echocardiogram, Holter ECG

Visit 7 (week 26+ 1 day): Hyperinsulinemic euglycemic clamp combined with 18F-FDG PET (shift of the treatment groups).

Visit 8 (week 30): Clinical examination, security monitoring (systolic and diastolic blood pressure), hypoglycemia and adverse events evaluation

Visit 9 (week 34): Clinical examination, security monitoring (ECG, blood pressure), hypoglycemia and adverse events evaluation

Visit 10 (week 40): Clinical examination, security monitoring, hypoglycemia and adverse events evaluation

Visit 11 (week 52): Clinical examination, vital signs, anthropometric measures, haematology and biochemistry, pro-BNP, high sensitivity C-reactive protein (hsCRP), troponin T, renal function, ACR, ECG, echocardiogram, Holter ECG.

Visit 12 (week 52 + 1 day): Hyperinsulinemic euglycemic clamp combined with 18F-FDG PET

Hyperinsulinemic euglycemic clamp combined with 18F-FDG-PET scan for assessment of peripheral insulin sensitivity and myocardial glucose uptake.

Myocardial metabolic rate of glucose (Global MRGlu - mmol/min/100mg) will be measured by 18F-FDG-PET acquired in the course of euglycemic hyperinsulinemic clamp as previously described. Subjects will be received a priming dose of insulin (Humulin R 100UI/ml; Eli Lilly) during the initial 10 min to acutely raise the desired levels of plasma insulin, followed by continuous insulin infusion fixed at 40 mU/m2 x min. The blood glucose level will be maintained constant at 90 mg/dl for the next 120 min by infusing 20% glucose at varying rates according to blood glucose measurements performed at 5-min intervals (mean coefficient of variation of blood glucose was <4%). Glucose metabolized by the whole body (M) will be calculated as the mean rate of glucose infusion measured during the last 60 minutes of the clamp examination (steady state) and was expressed as milligrams per minute per kilogram fat-free mass (MFFM).

The 18F-FDG PET imaging procedure will be performed on a hybrid PET/CT scanner (GE Discovery ST8- 2D PET scanner), starting 60 minutes after the insulin infusion. 60-min dynamic acquisition will be started simultaneously with the intravenous injection of 370 MBq18F-FDG and the insulin-glucose infusion will be continued during entire PET acquisition. The estimation of myocardial MRGlu will be performed using a Patlak compartmental modelling, a widely diffuse technique provided by a graphical tool specific for cardiac images analysis (PCARD) in PMOD Software platform (Version 3.806). PCARD allows to measure the global MRGlu as well as the segmental myocardial glucose uptake by using a segmentation algorithm to divide myocardium into standard 17 segments model according to ASNC (American Society of Nuclear Cardiology) guideline and the American Heart Association (AHA).

Sample size

The "Sample Size" in the study is of 26 subjects (13 subjects per group). The same result has been calculated considering a significant reduction in group Empagliflozin of 40 % in myocardial metabolic rate of glucose estimated through 18F-FGD-PET, compared to a change in the treatment arm glimepiride of 15% and assuming a standard deviation of 5%, a "dropout" of 10%, with a power of 85% and an alpha error of 0.05%, using the power calculation available at the following website https://clincalc.com/Stats/SampleSize.aspx.

The randomization of the subjects will be done using the program "Research Randomizer (www.randomizer.org). The subjects will be allocated to one of two arms of the study (1 = Treatment Empagliflozin; 2 = Treatment Glimepriride;) according to the outline generated by the program indicated above and attached to the protocol.

Safety assessment

During the course of the present study all adverse events (including hypoglycemic episodes), both those suspected to be study drug-related and those not suspected to be related to study medications, will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes, in treatment with metformin
* Written informed consent

Exclusion Criteria:

* Type 1 diabetes
* eGFR <60 ml/min/1.73 m2. or dialysis patients
* HbA1c <6.5 o >9%
* Previous treatment with insulin (except for short-term treatment with insulin in connection with intercurrent illness, at the discretion of the Investigator), with SGLT2 inhibitors or with GLP-1R agonists or DPPIV inhibitors
* Patients who do not tolerate empagliflozin and/or glimepiride or in whom empagliflozin and/or glimepiride are contraindicated
* Uncontrolled hypertension (BP>140/90 mmHg)
* Prior cardio- cerebral-vascular events
* Hepatic disease
* Pathology neoplastic (past or present)
* Pregnancy women or childbearing female without adequate and approved birth control method

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2021-10 (Actual); Study Completion 2021-10 (Actual)

PRIMARY OUTCOMES:
Change of myocardial metabolic rate of glucose | Baseline, after 26 and 52 weeks
  To assess whether empagliflozin treatment is able to determine a change of myocardial metabolic rate of glucose estimated through hyperinsulinemic euglycemic clamp 18FDG-PET scan, than glimepiride treatment (both in addition to metformin), in patients with T2DM without a history of coronary heart disease.

SECONDARY OUTCOMES:
Change of glycemic parameters | Baseline, after 26 and 52 weeks
  To compare empagliflozin and glimepiride (in addition to metformin) on glycemic parameters (fasting glucose, HbA1c).
Change of insulin sensitivity | Baseline, after 26 and 52 weeks
  To compare empagliflozin and glimepiride regimens on change of insulin sensitivity, assessed by hyperinsulinemic euglycemic clamp.
Change of blood pressure | Baseline, after 26 and 52 weeks
  To compare the respective impact of empagliflozin and glimepiride on systolic and diastolic blood pressure assessed at baseline and after 26 weeks
Change of left ventricular systolic and diastolic function | Baseline, after 26 and 52 weeks
  To compare empagliflozin and glimepiride on change of left ventricular systolic and diastolic function, assessed by echocardiogram
Change of pro-BNP | Baseline, after 26 and 52 weeks
  To compare the respective impact of empagliflozin and glimepiride on pro-BNP
Change of inflammatory state | Baseline, after 26 and 52 weeks
  To compare the respective impact of empagliflozin and glimepiride on high sensitivity C-reactive protein [hsCRP)
Change of cardiovascular biomarkers | Baseline, after 26 and 52 weeks
  To compare the respective impact of empagliflozin and glimepiride on cardiovascular biomarkers (troponin T)
Change of heart rate variability | Baseline, after 26 and 52 weeks
  To compare empagliflozin and glimepiride on change of heart rate variability assessed by Holter ECG
Change of lipid profile | Baseline, after 26 and 52 weeks
  To compare the respective impact of empagliflozin and glimepiride on lipid profile (total cholesterol, LDL cholesterol, HDL cholesterol, triglycerides)

CONTACTS AND LOCATIONS:
Overall Officials: Giorgio Sesti, MD, Study Director — University Sapienza of Rome
Locations (1):
- Universital Hospital Mater Domini, Catanzaro, Italy

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication. De-identified individual participant data for all primary and secondary outcomes will be made available
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Beginning 6 months and ending 36 months following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal. Proposals should be directed to succurro@unicz.it. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Background] Cho NH, Shaw JE, Karuranga S, Huang Y, da Rocha Fernandes JD, Ohlrogge AW, Malanda B. IDF Diabetes Atlas: Global estimates of diabetes prevalence for 2017 and projections for 2045. Diabetes Res Clin Pract. 2018 Apr;138:271-281. doi: 10.1016/j.diabres.2018.02.023. Epub 2018 Feb 26. PMID 29496507
- [Background] Vaccaro O, Eberly LE, Neaton JD, Yang L, Riccardi G, Stamler J; Multiple Risk Factor Intervention Trial Research Group. Impact of diabetes and previous myocardial infarction on long-term survival: 25-year mortality follow-up of primary screenees of the Multiple Risk Factor Intervention Trial. Arch Intern Med. 2004 Jul 12;164(13):1438-43. doi: 10.1001/archinte.164.13.1438. PMID 15249353
- [Background] Haffner SM, Lehto S, Ronnemaa T, Pyorala K, Laakso M. Mortality from coronary heart disease in subjects with type 2 diabetes and in nondiabetic subjects with and without prior myocardial infarction. N Engl J Med. 1998 Jul 23;339(4):229-34. doi: 10.1056/NEJM199807233390404. PMID 9673301
- [Background] Kannel WB, McGee DL. Diabetes and cardiovascular risk factors: the Framingham study. Circulation. 1979 Jan;59(1):8-13. doi: 10.1161/01.cir.59.1.8. PMID 758126
- [Background] Diabetes Control and Complications Trial Research Group; Nathan DM, Genuth S, Lachin J, Cleary P, Crofford O, Davis M, Rand L, Siebert C. The effect of intensive treatment of diabetes on the development and progression of long-term complications in insulin-dependent diabetes mellitus. N Engl J Med. 1993 Sep 30;329(14):977-86. doi: 10.1056/NEJM199309303291401. PMID 8366922
- [Background] Intensive blood-glucose control with sulphonylureas or insulin compared with conventional treatment and risk of complications in patients with type 2 diabetes (UKPDS 33). UK Prospective Diabetes Study (UKPDS) Group. Lancet. 1998 Sep 12;352(9131):837-53. PMID 9742976
- [Background] Green JB, Bethel MA, Armstrong PW, Buse JB, Engel SS, Garg J, Josse R, Kaufman KD, Koglin J, Korn S, Lachin JM, McGuire DK, Pencina MJ, Standl E, Stein PP, Suryawanshi S, Van de Werf F, Peterson ED, Holman RR; TECOS Study Group. Effect of Sitagliptin on Cardiovascular Outcomes in Type 2 Diabetes. N Engl J Med. 2015 Jul 16;373(3):232-42. doi: 10.1056/NEJMoa1501352. Epub 2015 Jun 8. PMID 26052984
- [Background] Udell JA, Cavender MA, Bhatt DL, Chatterjee S, Farkouh ME, Scirica BM. Glucose-lowering drugs or strategies and cardiovascular outcomes in patients with or at risk for type 2 diabetes: a meta-analysis of randomised controlled trials. Lancet Diabetes Endocrinol. 2015 May;3(5):356-66. doi: 10.1016/S2213-8587(15)00044-3. Epub 2015 Mar 17. PMID 25791290
- [Background] Standards of medical care in diabetes--2015: summary of revisions. Diabetes Care. 2015 Jan;38 Suppl:S4. doi: 10.2337/dc15-S003. No abstract available. PMID 25537706
- [Background] Abdul-Ghani MA, Norton L, Defronzo RA. Role of sodium-glucose cotransporter 2 (SGLT 2) inhibitors in the treatment of type 2 diabetes. Endocr Rev. 2011 Aug;32(4):515-31. doi: 10.1210/er.2010-0029. Epub 2011 May 23. PMID 21606218
- [Background] Ferrannini E, Muscelli E, Frascerra S, Baldi S, Mari A, Heise T, Broedl UC, Woerle HJ. Metabolic response to sodium-glucose cotransporter 2 inhibition in type 2 diabetic patients. J Clin Invest. 2014 Feb;124(2):499-508. doi: 10.1172/JCI72227. Epub 2014 Jan 27. PMID 24463454
- [Background] Zinman B, Wanner C, Lachin JM, Fitchett D, Bluhmki E, Hantel S, Mattheus M, Devins T, Johansen OE, Woerle HJ, Broedl UC, Inzucchi SE; EMPA-REG OUTCOME Investigators. Empagliflozin, Cardiovascular Outcomes, and Mortality in Type 2 Diabetes. N Engl J Med. 2015 Nov 26;373(22):2117-28. doi: 10.1056/NEJMoa1504720. Epub 2015 Sep 17. PMID 26378978
- [Background] Chilton R, Tikkanen I, Cannon CP, Crowe S, Woerle HJ, Broedl UC, Johansen OE. Effects of empagliflozin on blood pressure and markers of arterial stiffness and vascular resistance in patients with type 2 diabetes. Diabetes Obes Metab. 2015 Dec;17(12):1180-93. doi: 10.1111/dom.12572. Epub 2015 Oct 9. PMID 26343814
- [Background] Tikkanen I, Narko K, Zeller C, Green A, Salsali A, Broedl UC, Woerle HJ; EMPA-REG BP Investigators. Empagliflozin reduces blood pressure in patients with type 2 diabetes and hypertension. Diabetes Care. 2015 Mar;38(3):420-8. doi: 10.2337/dc14-1096. Epub 2014 Sep 30. PMID 25271206
- [Background] Rosenstock J, Jelaska A, Frappin G, Salsali A, Kim G, Woerle HJ, Broedl UC; EMPA-REG MDI Trial Investigators. Improved glucose control with weight loss, lower insulin doses, and no increased hypoglycemia with empagliflozin added to titrated multiple daily injections of insulin in obese inadequately controlled type 2 diabetes. Diabetes Care. 2014 Jul;37(7):1815-23. doi: 10.2337/dc13-3055. Epub 2014 Jun 14. PMID 24929430
- [Background] Santos-Gallego CG, Requena-Ibanez JA, San Antonio R, Ishikawa K, Watanabe S, Picatoste B, Flores E, Garcia-Ropero A, Sanz J, Hajjar RJ, Fuster V, Badimon JJ. Empagliflozin Ameliorates Adverse Left Ventricular Remodeling in Nondiabetic Heart Failure by Enhancing Myocardial Energetics. J Am Coll Cardiol. 2019 Apr 23;73(15):1931-1944. doi: 10.1016/j.jacc.2019.01.056. PMID 30999996
- [Background] Iozzo P, Chareonthaitawee P, Dutka D, Betteridge DJ, Ferrannini E, Camici PG. Independent association of type 2 diabetes and coronary artery disease with myocardial insulin resistance. Diabetes. 2002 Oct;51(10):3020-4. doi: 10.2337/diabetes.51.10.3020. PMID 12351442
- [Background] Nishikawa J, Ohtake T, Yokoyama I, Watanabe T, Momose T, Sasaki Y. Simple method to quantify myocardial glucose metabolism from MB ratio in myocardial FDG PET. Ann Nucl Med. 1996 Aug;10(3):323-8. doi: 10.1007/BF03164739. PMID 8883708
- [Background] Gerber BL, Ordoubadi FF, Wijns W, Vanoverschelde JL, Knuuti MJ, Janier M, Melon P, Blanksma PK, Bol A, Bax JJ, Melin JA, Camici PG. Positron emission tomography using(18)F-fluoro-deoxyglucose and euglycaemic hyperinsulinaemic glucose clamp: optimal criteria for the prediction of recovery of post-ischaemic left ventricular dysfunction. Results from the European Community Concerted Action Multicenter study on use of(18)F-fluoro-deoxyglucose Positron Emission Tomography for the Detection of Myocardial Viability. Eur Heart J. 2001 Sep;22(18):1691-701. doi: 10.1053/euhj.2000.2585. PMID 11511119
- [Background] Marini MA, Succurro E, Frontoni S, Mastroianni S, Arturi F, Sciacqua A, Lauro R, Hribal ML, Perticone F, Sesti G. Insulin sensitivity, beta-cell function, and incretin effect in individuals with elevated 1-hour postload plasma glucose levels. Diabetes Care. 2012 Apr;35(4):868-72. doi: 10.2337/dc11-2181. Epub 2012 Feb 22. PMID 22357182
- [Background] Morbelli S, Marini C, Adami GF, Kudomi N, Camerini G, Iozzo P, Massollo M, Capitanio S, Bodrato S, Verardi MT, Papadia F, Cordera R, Knuuti J, Scopinaro N, Sambuceti G. Tissue specificity in fasting glucose utilization in slightly obese diabetic patients submitted to bariatric surgery. Obesity (Silver Spring). 2013 Mar;21(3):E175-81. doi: 10.1002/oby.20003. PMID 23404920
- [Background] Cerqueira MD, Weissman NJ, Dilsizian V, Jacobs AK, Kaul S, Laskey WK, Pennell DJ, Rumberger JA, Ryan T, Verani MS; American Heart Association Writing Group on Myocardial Segmentation and Registration for Cardiac Imaging. Standardized myocardial segmentation and nomenclature for tomographic imaging of the heart. A statement for healthcare professionals from the Cardiac Imaging Committee of the Council on Clinical Cardiology of the American Heart Association. Circulation. 2002 Jan 29;105(4):539-42. doi: 10.1161/hc0402.102975. No abstract available. PMID 11815441